CLINICAL TRIAL: NCT03295942
Title: A Phase 1a Open-Label, Dose Escalation Study of the Safety and Pharmacokinetics of OMP-336B11 Administered as a Single Agent to Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of OMP-336B11 in Subjects With Locally Advanced or Metastatic Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 336B11-001
Record Dates: First submitted 2017-09-13; First posted 2017-09-28 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Locally Advanced Malignant Neoplasm; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: OMP-336B11
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OMP-336B11 (Experimental): Intravenous (in the vein) infusions of OMP-336B11
  Interventions: Drug: OMP-336B11

INTERVENTIONS:
Drug: OMP-336B11 — OMP-336B11 is an engineered human protein that was designed to bind to the GITR receptor on T cells and activate the immune system to recognize and eliminate cancer cells.

SUMMARY:
The purpose of this study is to test the safety and efficacy of OMP-336B11. OMP-336B11 is an engineered human protein that was designed to bind to the GITR receptor on T cells and activate the immune system to recognize and eliminate cancer cells.

DETAILED DESCRIPTION:
This is an open-label, Phase 1a dose escalation study of OMP-336B11 administered as a single agent to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics in patients with locally advanced or metastatic tumors. This study consists of a screening period, a treatment period, and a post-treatment follow-up period in which patients will be followed for survival for up to approximately 2 years. Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic solid tumors that have exhausted standard of care therapy
* Measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1
* Age >21 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and marrow function
* For women of childbearing potential and men with partners of childbearing potential, agreement (by patient and/or partner) to use two effective forms of contraception from study entry through at least 6 months after the termination visit.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Receiving any other investigational agents or any other anti-cancer therapy
* Active autoimmune disease or a history of severe autoimmune disease or syndrome
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Pregnancy, lactating or breastfeeding women
* History of primary CNS malignancy, or leptomeningeal disease or CNS metastases
* Significant uncontrolled intercurrent illness that will limit the patient's ability to participate in the study
* Inability to comply with study and follow up procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) or maximum administered dose (MAD) will be determined in patients treated with OMP-336B11 | Subjects will be assessed for DLTs through the end of the first cycle (Days 1-29)
  Incidence of dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Pharmacokinetic Outcome Measures (CL) | Screening through 12 weeks post treatment termination
  Clearance (CL) will be evaluated
Pharmacokinetic Outcome Measures (Vd) | Screening through 12 weeks post treatment termination
  Volume of distribution (Vd) will be evaluated
Pharmacokinetic Outcome Measures (T1/2) | Screening through 12 weeks post treatment termination
  The half life (T1/2) of OMP-336B11 will be assessed
Immunogenicity of OMP-336B11 (Percentage of patients with anti-336B11 antibodies) | up to approximately 2 years
  Percentage of patients with anti-336B11 antibodies assessed
Objective Response | up to approximately 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Progression-Free Survival | up to approximately 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos P Papadopoulos, MD, Principal Investigator — South Texas Accelerated Research Therapeutics, LLC
Locations (1):
- South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No